CLINICAL TRIAL: NCT01270191
Title: The Effects of Short-Term Exenatide Therapy on the Beta-Cell Function and Long-term Glycemic Control in Newly Diagnosed Type 2 Diabetic Patients
Brief Title: The Effects of Short-Term Exenatide Therapy in Newly Diagnosed Type 2 Diabetic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Taipei Veterans General Hospital, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHIRB 201010013MB
Record Dates: First submitted 2011-01-03; First posted 2011-01-05 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Type 2 Diabetes
Keywords: Exenatide, Beta-Cell Function, Glycemic Control; in Newly Diagnosed Type 2 Diabetic Patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Experimental): In the exenatide therapy group, subjects will be instructed in the techniques for injection and be treated with 5 mcg bid for 4 weeks and then 10 mcg bid for 12 weeks. They also visit every 2 weeks in the first 2 visits and then every month until 4 months. If FPG still greater than 200 mg/dL after 4 weeks of exenatide treatment, they will use insulin for rescue therapy and will be withdrawn from this study.
  Interventions: Drug: Exenatide
- Humulin-N (Active Comparator): In the insulin therapy group (Humulin-N), subjects will be instructed in the techniques for insulin injection and home capillary glucose monitoring. The insulin dose will be initiated with 0.25 unit/Kg per day, and the two thirds of daily dose will be administrated before breakfast and the other will be administrated at bedtime. Insulin doses will be titrated every 3 days to achieve target fasting blood glucose values between 70 and 130 mg/dl.
  Interventions: Drug: Humulin-N

INTERVENTIONS:
Drug: Exenatide — They will be treated with 5 mcg bid for 4 weeks and then 10 mcg bid for 12 weeks. They also visit every 2 weeks in the first 2 visits and then every month until 4 months.
  Other Names: Byetta
  Arms: Exenatide
Drug: Humulin-N — The insulin dose will be initiated with 0.25 unit/Kg per day, and the two thirds of daily dose will be administrated before breakfast and the other will be administrated at bedtime. Insulin doses will be titrated every 3 days to achieve target fasting blood glucose values between 70 and 130 mg/dl.
  Other Names: NPH insulin
  Arms: Humulin-N

SUMMARY:
Whether GLP-1 and GLP-1 receptor agonists will produce a sustained improvement in beta-cell function following short-term therapy is currently not known. This randomized, controlled trial is carried to assess the efficacy of short-term insulin therapy (NPH injection twice daily) compared with GLP-1 analogue (Exenatide injection twice daily) on glycemic control, remission rate, ß-cell function, and long-term glycemic control in newly diagnosed type 2 diabetic patients with moderate hyperglycemia.

DETAILED DESCRIPTION:
Background: There is a progressive deterioration in beta-cell function in type 2 diabetics, and it was estimated that islet function was about 50% of normal at the time of diagnosis. The progressive nature of type 2 diabetes is one of the major challenges in the treatment of affected patients, and agents that could alter the natural history of this condition would add greatly to current treatment approaches. Short-term intensive insulin therapy of newly diagnosed type 2 diabetes will improve beta-cell function and usually leading to a temporary remission time. The acute effect of GLP-1 and GLP-1 receptor agonists on beta-cells is stimulation of glucose-dependent insulin release, followed by enhancement of insulin biosynthesis and stimulation of insulin gene transcription. The chronic action is stimulating beta-cell proliferation, induction of islet neogenesis, and inhibition of ß-cell apoptosis, thus promoting expansion of beta-cell mass, as observed in rodent diabetes and in cultured beta-cells.

Objectives: Whether GLP-1 and GLP-1 receptor agonists will produce a sustained improvement in beta-cell function following short-term therapy is currently not known. This randomized, controlled trial is carried to assess the efficacy of short-term insulin therapy (NPH injection twice daily) compared with GLP-1 analogue (Exenatide injection twice daily) on glycemic control, remission rate, beta-cell function, and long-term glycemic control in newly diagnosed type 2 diabetic patients with moderate hyperglycemia.

Study Designs and Methods: We will recruit 80 newly diagnosed type 2 diabetic patients with moderate hyperglycemia, and another 80 newly diagnosed type 2 diabetic patients with severe hyperglycemia who receive intensive insulin therapy for 10-14 days, and will be randomized to be treated with exenatide or insulin injections. They will visit our clinics every 2 weeks in the first 2 visits and then every 4 weeks for 20 weeks. After the 24 weeks of intervention, all patients will be treated with life style modification only and follow fasting plasma glucose every month. Hyperglycemia relapse is defined as fasting plasma glucose more than 126 mg/dL and confirmed two weeks later. Patients with hyperglycemia relapse will be treated with metformin (from 500 mg per day to 1500 mg per day)and then gliclazide-MR will be added to as the second step for the remaining study period. A1C measurement will be performed at baseline, 3, 6, 12 and 18 months, and OGTT will be performed at screen and after 6 months of randomization. All of these subjects were continually followed-up in our clinics for 5 years to evaluate their long-term glycemic control. The monotherapy failure is defined as A1C >7.0% with metformin 1500 mg/day.

The primary outcomes at one year are the time of glycemic remission and remission rate at one year after short-term therapy. The primary outcomes at 5 years are monotherapy failure time and monotherapy failure rate at 5 years after short-term therapy. The secondary outcomes are the beta-cell function and insulin sensitivity calculated from OGTT, the comparison of A1C change, the proportion of subjects who reached the treatment target (A1C <7.0% or <6.5% at 1 and 5 years). These subjects will be followed up for 5 years to evaluate their long-term glycemic control.

Expected Results: We will expect to screen 100 patients, randomize 80 patients and there will be at least 30 patients in each group complete the one year follow-up. We expected that short-term intensive treated with both insulin and exenatide can get better glycemic control accompanied with improving the beta-cell function in newly diagnosed type 2 diabetes. We can compare the remission rate at one year after different short-term therapy. We will further evaluate the effects on the beta-cell function and long-term glycemic control. This study also can assess what readily available parameter would predict which patients will achieve long-term successful glycemic control after correction of glucose toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed type 2 diabetic patients.
2. Age between 30 and 70 years old.
3. HbA1C between 7 and 9% in OPD patients
4. If HbA1c >9.0% of blood glucose >300 mg/dL, intensive insulin therapy for 10-14 days

Exclusion Criteria:

1. Previous treated with anti-diabetic medication
2. Pregnant or lactation women.
3. Impaired liver function (ALT > 100 U/L)
4. Impaired renal function (Serum creatinine >2.0 mg/dL)
5. Recently suffered from MI or CVA.
6. Patients are acute intercurrent illness.
7. 2-hour C-peptide level < 2.0 ng/mL.
8. History of severe hypersensitivity to any product components.
9. History or high risk of acute pancreatitis.
10. Now use warfarin.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-11; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
the time of glycemic remission and remission rate | at one year
  The primary outcomes are the time of glycemic remission and remission rate at one year after short-term therapy.
The time of monotherapy failure and monotherapy failure rate | 5 years
  The primary outcomes at 5 years are long-term glycemic control. After 5 months of intensive therapy, these patients were off medication and follow up in our clinics. When diabetes relapsed, they will be treated with metformin monotherapy. The monotherapy failure is defined as A1C >7.0% with metformin 1500 mg per day.

SECONDARY OUTCOMES:
Beta-cell function and insulin sensitivity calculated from OGTT. | at 6 months
  The Beta-cell function and insulin sensitivity calculated from OGTT.
Comparison of A1C change, the proportion of subjects who reached the treatment target | 6-12 months
  The secondary outcomes are the comparison of A1C change, the proportion of subjects who reached the treatment target (A1C <7.0% or <6.5%) at 6 months and 12 months.
Comparison of A1C change, the proportion of subjects who reached the treatment target | 5 years
  These subjects will be followed up for 5 years to evaluate their long-term glycemic control. The secondary outcomes are the comparison of A1C change, the proportion of subjects who reached the treatment target (A1C <7.0% or <6.5%) at 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Harn-Shen Chen, MD, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taipei, Taiwan